CLINICAL TRIAL: NCT05502068
Title: A Randomized, Placebo-controlled, Independent Study of the Positive, Quantifiable Effects of Sublingual Spray LYL Love Your Life® sunD3 LYLmicro™ (LYLmicro™) on Blood Levels of Vitamin D3 and Inflammatory Markers in Patients With COVID-19
Brief Title: The Effects of a Sublingual Sprayable Microemulsion of Vitamin D on Inflammatory Markers in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021sunD3LYLmicroTMSARS-CoV-2
Record Dates: First submitted 2022-08-15; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; Vitamin D Deficiency
Keywords: COVID-19; CRP; Vitamin D insufficiency; Vitamin D spray
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency | interventions — hydroxide ion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D 25 (OH) 12000 IU, Sublingual sprayable microemulsion (Experimental): Vitamin D in the form of a sublingual sprayable microemulsion (4000 IU) will be given three times daily after breakfast, lunch, and dinner (daily dose 12,000 IU) to patients with blood vitamin D levels below 30 ng/ml for 5-day intervention
  Interventions: Dietary Supplement: Vitamin D 25 (OH) 12000 IU in the form of a sublingual sprayable microemulsion
- Placebo (Placebo Comparator): Placebo will be given to the control group. It will be administrated sublingually, with one spray three times per day for 5 days of the study period
  Interventions: Dietary Supplement: Vitamin D 25 (OH) 12000 IU in the form of a sublingual sprayable microemulsion

INTERVENTIONS:
Dietary Supplement: Vitamin D 25 (OH) 12000 IU in the form of a sublingual sprayable microemulsion — This is a prospective, randomized, double blind, and controlled clinical study to investigate the impact of the high dose vitamin D supplementation on laboratory markers of systemic inflammation such as CRP, ferritin and IL-6 in hospitalized patients with COVID-19. Patients included in the study will be randomized into two groups and receive a placebo (as a control group) or cholecalciferol administered sublingually for 5 day

SUMMARY:
This placebo-controlled five-day study will be performed on 100 hospitalized COVID-19 patients with vitamin D insufficiency randomized into two groups. Vitamin D in the form of a sublingual sprayable microemulsion (LYL love your life® sunD3 LYLmicro™) is given three times daily after breakfast, lunch, and dinner (daily dose 12,000 IU) to patients with blood vitamin D levels below 30 ng/ml. The control (placebo) group recieves a placebo spray in the same daily regimen.

DETAILED DESCRIPTION:
This placebo-controlled five-day study will be performed on 100 hospitalized COVID-19 patients with vitamin D insufficiency randomized into two groups.

The aim of this study is to investigate the impact of the high dose vitamin D supplementation on laboratory markers of systemic inflammation such as CRP, ferritin and IL-6 in hospitalized patients with COVID-19. The blood samples are analyzed at the Joint Laboratory of the Pauls Stradins Clinical Univesity Hospital. Patients with confirmed SARS-CoV2 infection (PCR) will be randomly divided into two groups: the intervention group receives vitamin D in the form of a sublingual sprayable microemulsion (LYL love your life® sunD3 LYLmicro™) of 4,000 IU three times daily after breakfast, lunch and dinner; the control group receives the same regimen of placebo spray.

A total of 100 inpatients will be selected for the study. All patients will receive standard care for COVID-19 and existing comorbidities (diabetes, arterial hypertension, etc) according to hospital-approved protocol. The primary outcome is defined as the change in the level of the inflammatory marker and the disease's severity.

Population. Disease severity is defined by the blood oxygen saturation level. Mild clinical manifestation is characterized by SpO2≥94%, moderate 90%≤SpO2<94% and severe - SpO2<90%. Age, BMI, GFR, vitamin D and COVID-19 severity are considered as randomization parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 and over
* Vitamin D level below 30 ng/ml
* Positive SARS-CoV-2 test

Exclusion Criteria:

* Patients with mental health problems,
* eGFR ≤30 ml/min,
* Vitamin D level ≥ 30 ng/ml,
* Pregnant women
* Any other illness or condition that the researcher deemed may interfere with the results
* Patients who refuse the studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Evaluating the effects of a sprayable microemulsion of cholecalciferol on vitamin D levels in the blood of COVID-19 patients | month 1-4
  The study's primary outcome is to demonstrate the efficacy of sprayable microemulsion of cholecalciferol on the increase in circulating vitamin D levels over a period of at least 5 days.

SECONDARY OUTCOMES:
Evaluating the effects of a sprayable microemulsion of cholecalciferol on inflammatory markers in the blood of COVID-19 patients | Month 1-4
  The study's secondary outcome is to demonstrate the efficacy of sprayable microemulsion of cholecalciferol on inflammatory markers (blood cell count, CRP, fibrinogen, IL-6) in COVID-19 patients with vitamin D levels below 29.9 ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Valdis Pirags, MD, PhD, Principal Investigator — Pauls Stradins Clinical University Hospital
Locations (1):
- Pauls Stradins Clinical Univeristy Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No